CLINICAL TRIAL: NCT01501630
Title: Role of PET/CT With Fluorine-18 Tracers and of Diffusion Weighted Whole-body MRI in the Early Detection of Bone Metastases in Prostate Cancer
Brief Title: Role of PET/CT With Fluorine-18 Tracers of Bone Metastases in Prostate Cancer
Acronym: FLUPROSTIC
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P090105; 2011-A01041-40 (Other: IDRCB)
Record Dates: First submitted 2011-12-26; First posted 2011-12-29 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: Comparison of imaging modalities; Impact on patient management; Optimisation of cost of the diagnostic strategy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PET/CT and MRI: all patients will benefit from PET/CT and MRI
  Interventions: Device: performance of PET/CT and whole-body MRI

INTERVENTIONS:
Device: performance of PET/CT and whole-body MRI — For PET/CT radiopharmaceuticals, both registered in France:Fluoride (18F)FLUOROCHOLINE (18F)No contrast agent scheduled for MRI in the study RadiopharmaceuticalsSingle use, 2-4 MBq/kg body weight, IV infusion

SUMMARY:
Compare PET/CT and MRI for the early detection of bone metastases of prostate cancer: diagnostic performance and impact on the patient management.Determine the lowest cost strategy according to the precise clinical circumstances.

DETAILED DESCRIPTION:
In patients with high risk prostate cancer and high PSA levels, PET/CT with fluoride (18F) and FLUOROCHOLINE (18F) and whole-body MRI will be performed within one month.

Data of a 6 month follow-up after those examination will be made available to a panel of independent experts. They will determine the standard of truth (SOT) concerning the invasion of the skeleton and also of soft tissue by prostate cancer tissue, the impact of each imaging modality on patient management and the adequacy of the decisions. In some cases (anti-hormone treatment without histology), it will not be possible to determine the SOT.

By comparison of the results of blind readings for each imaging modality with the standard of truth, the diagnostic performance will be determined.

By simulation, several strategies will be constructed concerning the best examinations to be performed and the sequence according to the precise clinical circumstances. Their cost and effectiveness will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Histologically proven prostate cancer.
* Abnormal plasmatic level of prostate specific antigen dating less than 3 months, initial Gleason score available
* Written informed consent.

Exclusion Criteria:

* Other active cancer or bone infection.
* Chemotherapy or change in hormone therapy since the last PSA assay
* Contraindication to MRI without contrast agent (claustrophobia, pace maker, metallic foreign body, some cardiac valves). Metallic joint prostheses are NOT a contraindication.
* Allergic reaction to radiopharmaceuticals that will be used.
* Patient who seems not capable of staying in the gantry of the machines during the examinations without moving.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
bone metastases | within 6 months
  Follow up data (histology, imaging, PSA levels) during 6 months to determine the standard of truth and the adequacy of the management decided on basis of imaging modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Noël TALBOT, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service Médecine Nucléaire - Hôpital TENON, Paris, France

REFERENCES:
- [Derived] Gauthe M, Zarca K, Aveline C, Lecouvet F, Balogova S, Cussenot O, Talbot JN, Durand-Zaleski I. Comparison of 18F-sodium fluoride PET/CT, 18F-fluorocholine PET/CT and diffusion-weighted MRI for the detection of bone metastases in recurrent prostate cancer: a cost-effectiveness analysis in France. BMC Med Imaging. 2020 Mar 2;20(1):25. doi: 10.1186/s12880-020-00425-y. PMID 32122345